CLINICAL TRIAL: NCT04544540
Title: One Versus Two Unit Transfusions in Oncology Patients - The OTTOP Trial: A Randomized Open-label Pragmatic Controlled Trial
Acronym: OTTOP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20200578-01H
Record Dates: First submitted 2020-09-04; First posted 2020-09-10 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Anemia; Oncology
MeSH Terms: conditions — Anemia; Neoplasms

STUDY DESIGN:
Intervention Model Description: A randomized open-label pragmatic controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- One-Unit (Experimental): Patients will be randomized to receive 1-unit of red blood cell transfusions as an outpatient a period of one-year. At each outpatient transfusion episode, the patient will receive a transfusion of 1-unit
  Interventions: Other: Units of transfusion
- Two-Unit (Experimental): Patients will be randomized to receive 2-unit sof red blood cell transfusions as an outpatient a period of one-year. At each outpatient transfusion episode, the patient will receive a transfusion of 2-units
  Interventions: Other: Units of transfusion

INTERVENTIONS:
Other: Units of transfusion — Participants will either receive 1-unit or 2-unit red blood cell outpatient transfusions

SUMMARY:
The aim of this trial is to determine if the transfusion of one unit of red blood cells to anemic oncology patients results in comparable numbers of transfusion episodes when compared to transfusion of two units of red blood cells.

DETAILED DESCRIPTION:
The aim of this trial is to determine if administration of one unit of red blood cells to anemic oncology patients is non-inferior to the administration of two units of red blood cells in terms of the number of annual transfusion episodes. If demonstrated, our findings will cut the total transfusion episode time in half and avoid exposure to an additional unit of red blood cells while freeing up scarce hospital resources.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 18 years of age with solid tumour (non-hematologic) malignancy undergoing chemotherapy
* Requiring a red blood cell transfusion as determined by their treating oncologist

Exclusion Criteria:

* Active bleeding (WHO grade 3 and 4)
* Known history active hemolysis
* Inpatient admission
* Refusal to receive red blood cell transfusion
* Unwilling or unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2023-11-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
number of transfusion episodes in the 1-year after randomization | 1 year

SECONDARY OUTCOMES:
Total number of transfusion episodes per patients per month while on chemotherapy. | 1 year
Total number of units transfused while on chemotherapy and for entire 1-year follow-up | 1 year
Duration of outpatient transfusion episodes (time in the medical day care unit) | 1 year
Hemoglobin levels at the time of next (1st post transfusion) chemotherapy treatment. | 1 year
Hemoglobin levels at the time of subsequent chemotherapy treatments | 1 year
Post-transfusion hemoglobin increment defined as the difference between the pretransfusion and first hemoglobin measurement occurring after the completion of the transfusion. | 1 year
The number of delays in any subsequent chemotherapy treatments. | 1 year
The length of delays in any subsequent chemotherapy treatments. | 1 year
Visits to the emergency department and hospitalizations. | 1 year
Difference in Pre- and post-transfusion Edmonton Symptom Assessment Scale where available | 1 year
Cancer status at 1- year post randomization | 1 year
Adverse transfusion reactions. | 1 year